CLINICAL TRIAL: NCT03185182
Title: "An Exploratory Study Regarding the Use of the Biomarker Dopamine Transporter (DAT) for Image Diagnosis of Clear Cell Renal Cell Carcinoma"
Brief Title: Diagnostic Imaging for Clear Cell Renal Cell Carcinoma
Acronym: RCCSCAN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to "early stopping rule" as defined in the study protocol
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RCCSCAN; 2016-005182-31 (EudraCT Number)
Record Dates: First submitted 2017-06-02; First posted 2017-06-14 (Actual); Results first posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-03

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: Diagnosis; Imaging
MeSH Terms: conditions — Carcinoma, Renal Cell; Disease | interventions — ioflupane

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental group (Experimental): 185 megabecquerel (MBq) of Ioflupane I-123 (DaTSCAN) will be administered IV to patients with suspected renal cell carcinoma, at a single occasion and followed by SPECT-analysis 5h after injection.The images from the DaTSCAN investigation will be analyzed and anatomically compared to CT-scan from the same the patient. Any adverse effects during the study will be reported.
  This is a exploratory open single arm trial, including a small number of patients with suspected disseminated renal cell carcinoma.
  Interventions: Drug: Ioflupane I123

INTERVENTIONS:
Drug: Ioflupane I123 — 185 MBq ioflupane I123 will be administered at one single occasion to the study subjects A one time dose of DaTSCAN is given via intravenous injection of 185 MBq Ioflupane (I123) .
  The patient takes potassium iodine tablets prior to the DatSCAN injection to protect the thyroid gland. At the time of the DaTSCAN examination, the patient is injected intravenously at slow rate with 185MBq DaTSCAN solution.
  Other Names: DaTSCAN

SUMMARY:
The main objective is to study whether imaging detection of the biomarker DAT can be used to detect kidney tumors identified by computer tomography (CT), which are pathologically assesses as being of the clear cell subtype.

DETAILED DESCRIPTION:
Main objective of the trial:

The main objective is to investigate whether DaTSCAN with subsequent SPECT can detect elevated DAT levels in at least a lesion identified with CT in patients with clear cell renal cell carcinoma, as assesed by pathologist? DaTSCAN signal will be seen as positive, displaying intensity ≥3ggr higher than the background and correlating anatomically with at least one lesion found with CT. DaTSCAN is used routinely to detect the loss of dopaminergic neurons in the striatum of patients with clinically uncertain Parkinsonian Syndromes. The active substance in DaTSCAN, Ioflupane specifically binds to DAT. By analyzing the focal uptake of Ioflupane (123I) with SPECT / CT the progression of the disease may be clarified. In light of our findings that clear cell renal cancer express significantly elevated levels of DAT, we postulate that DaTSCAN can be used for detection of clear cell renal cell carcinoma.

Protection of trial subjects:

Very few adverse effects are reported for DatSCAN use. In this study we used the same dose and route of administration as is praxis for DaTSCAN when used for diagnostic investigation of Parkinsons disease. Albeit uncommon, pain at the injection site has been previously reported when the solution was injected into a small vain. To minimise the potential for pain at the injection site during administration in this study, a slow intravenous injection (not less than 15 to 20 seconds) via an arm vein was therefore applied. The injections were performed by routined staff at Skåne University Hospital, Department of Clinical Physiology / Nuclear Medicine in Malmö, where usual clinical preparedness for allergic reactions after injection was available.

Background therapy:

Patients underwent appropriate thyroid blocking treatment prior to injection of DaTSCAN, to minimise thyroid uptake of radioactive iodine. In this study, this was achieved by oral administration of 2x 65 mg potassium iodide tablettes on the night before the DaTSCAN investigation and another 2x 65 mg potassium iodine tabletts 1 hour prior to injection of DaTSCAN.

ELIGIBILITY:
Inclusion Criteria:

* suspected kidney cancer diagnosis
* suspected spread of the cancer
* patient is scheduled for surgery alternatively biopsy of kidney tumor
* patient is 18 years or older
* the patient has given their consent to participate in the study
* female patients of reproductive age displays negative pregnancy test

Exclusion Criteria:

* known or suspected allergy to Ioflupane or sodium acetate or acetic acid or ethanol
* patient suffers from moderate to severe renal impairment and exhibits glomerular filtration rate (GFR) <40
* patient is medicated for Parkinson's disease
* patient is medicated with any of the following medications: amphetamine, benzatropine, buproprion, cocaine, mazindol, methylphenidate, phentermine, sertraline, levodopa, dexamphetamine, lisdexamphetamine, modafinil, moclobemid, venlafaxine
* patient is pregnant
* breastfeeding
* patient suffers from mental inability unwillingness or language difficulties resulting in difficulty in understanding the meaning of taking part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Elfving, M.D. PhD, Principal Investigator — Region Skane
Locations (1):
- Skåne University hospital SUS, Lund, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited continously in this study. Five patients were recruited, all at the Urological Clinic at Skåne University Hospital, Jan Waldenströms gata 7, 205 02 Malmö, Sweden. The first patient was recruited 2017-07-14 and the last patient was recruited at 2018-05-23.
Pre-assignment Details: Patients were recruited continously in this study. Screening critera: suspected dissiminated renal cancer, age 18-70. Five patients were screened for the study and all five patients were considered suitable for enrollment.
Groups:
- Experimental Group: 185 megabecquerel (MBq) of Ioflupane I-123 will be administered IV to patients with suspected renal cell carcinoma, at a single occasion and followed by SPECT-analysis 5h after injection.
  Ioflupane I123: 185 MBq ioflupane I133 will be administered at one single occasion to the study subjects
Period: Overall Study
Arm/Group | Experimental Group
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Group
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 55 [23 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 5
RCC subtype [Count of Participants; unit: Participants] — Pathological assessment of renal cell carcinoma (RCC) subtype was determined following surgical resection of the tumour. This occurs after DaTSCAN analysis.
  Classified as ccRCC=clear cell renal cell carcinoma or non-ccRCC=all other subtypes of kidney cancer
  Participants
    ccRCC | 4
    non-ccRCC | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Display Ioflupane-positivity in Tumors Detected Via CT-scan
Description: The primary endpoint is to investigate if tumors detected with CT display Ioflupane positivity in patients with verified clear cell renal cell carcinoma (ccRCC). Ioflupane signal was considered positive when intensity was >3 times background signal in anatomic position identified as a lesion by CT-scan
Time Frame: Through study completion for each participant, an average of 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Experimental Group: 185 megabecquerel (MBq) of Ioflupane I-123 will be administered IV to patients with suspected renal cell carcinoma, at a single occasion and followed by SPECT-analysis 5h after injection.
  Ioflupane I123: 185 MBq ioflupane I123 will be administered at one single occasion to the study subjects
Arm/Group | Experimental Group
Number analyzed (Participants) | 5
Participants | 0

2. Secondary Outcome: Number of Participants Diagnosed With Non-ccRCC That Display Ioflupane I123-negativity in Tumors Detected Via CT-scan
Description: Ioflupane I123 displays no positive signal in lesions identifies by CT in patients with tumors classified as non-clear cell renal cell carcinoma
Time Frame: Through study completion for each participant, an average of 3 months
Population: Patients with non-ccRCC as verified by pathologist
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: AE were reported consecutively for each patient while included in the trial, from potassium iodide intake to two days after Datscan examination, 4 days in total.
Description: AE were reported consecutively for each patient while included in the trial. Incidents may be observed by a doctor / nurse or reported by the subjects themselves. The subjects were asked an open question "Have you had any health problems since taking potassium iodide?" at each relevant study visit (below).
  * When injecting DaTSCAN (Ioflupan I123)
  * Immediately after the SPECT investigation
  * 2 days after the DaTSCAN examination (through telephone interview from research nurse)
Arm/Group | Experimental Group
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
Only 5 out of 10 intended patients were recruited in the study due to "early stopping rule" as defined in the study protocol as: terminate study if 4 patients with, by pathologist verified, ccRCC all display negative ioflupane signal in all lesions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT03185182/Prot_SAP_000.pdf